CLINICAL TRIAL: NCT02635802
Title: the Research of Analgesia and Sedation Effect of Remifentanil on ICU Short Operation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Principal Investigator, Rongqi Sun, The director of SICU,Chief physician,professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zdyfysicu-1
Record Dates: First submitted 2015-12-06; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Critical Illness
Keywords: remifentanil; analgesia; intensive care units
MeSH Terms: conditions — Critical Illness; Agnosia | interventions — Remifentanil; Lidocaine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Remifentanil (Experimental): injection form concentration 20μg/ml loading dose 1.0-2.0μg/kg intravenous injection slowly,time >1min,then 5μg/kg·h pumping until the operation is finished.
  Interventions: Drug: Remifentanil; Drug: Midazolam
- Lidocaine (Experimental): injection form concentration 10mg/ml loading dose 100-400mg local anesthesia
  Interventions: Drug: Lidocaine; Drug: Midazolam
- Remifentanil+Lidocaine (Experimental): injection form concentration 20μg/ml loading dose 1.0-2.0μg/kg intravenous injection slowly,time >1min,then 5μg/kg·h pumping until the operation is finished
  + injection form concentration 10mg/ml loading dose 100-400mg local anesthesia
  Interventions: Drug: Remifentanil+Lidocaine; Drug: Midazolam

INTERVENTIONS:
Drug: Remifentanil — a loading dose 1.0-2.0μg/kg remifentanil,intravenous injection slowly,time >1min,then 5μg/kg·h pumping if the operation can not be done in 5 minutes.
  Critical-Care Observation Tool(CPOT) and Richmond Agitation-Sedation Scale(RASS) are assessed before and after the loading.We should maintain the CPOT≤2 and RASS 0～2,if it is not up to the standard,increasing the pumping rate 0.5 μg/kg·h every 2-5min.
  Arms: Remifentanil
Drug: Lidocaine — lidocaine 100-400mg,local anesthesia.Critical-Care Observation Tool(CPOT) and Richmond Agitation-Sedation Scale(RASS) are assessed before and after local anesthesia.We should maintain the CPOT≤2 and RASS 0～2.
  Arms: Lidocaine
Drug: Remifentanil+Lidocaine — a loading dose 1.0-2.0μg/kg remifentanil,intravenous injection slowly,time >1min,then 5μg/kg·h remifentanil pumping immediately if the operation can not be done in 5 minutes.then local anesthesia with lidocaine 100-400mg.Critical-Care Observation Tool(CPOT) and Richmond Agitation-Sedation Scale(RASS) are assessed before and after anesthesia.We should maintain the CPOT≤2 and RASS 0～2,if it is not up to the standard,increasing the pumping rate 0.5μg/kg·h every 2-5min.
  Arms: Remifentanil+Lidocaine
Drug: Midazolam — midazolam is an adjuvant drug.we should maintain the CPOT≤2 and RASS 0～2,if lidocaine is already used up to 400mg or the pumping rate of remifentanil is already 7.5μg/kg·h,then we should use midazolam 3mg, intravenous injection slowly.

SUMMARY:
Remifentanil is one kind of opiates with strong analgesic effect,which has the rapid onset and short lasting duration. Remifentanil usually is used to help reducing the pain of patients with mechanical ventilation in ICU. Maybe it can also be used to ease the pain in ICU small short time operation.The purpose of this study is to determine (1) whether remifentanil is effective in small short time operations in ICU or not, (2) the save range of remifentanil in small short time operations in ICU, (3) and the adverse reaction that happens in these operations.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients need endotracheal intubation
* tracheotomy
* central venous puncture
* pleural puncture
* abdominal puncture
* lumbar puncture
* bone marrow puncture
* fiber bronchoscopic examination
* other small short-time operations

Exclusion Criteria:

* patients allergic to opioids
* in pregnancy or in feeding
* with myasthenia gravis
* with hypovolemia,
* take monoamine oxidase inhibitor(MAOI) in 14days
* in coma and GCS<8
* with bradycardia or hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
vital signs change | baseline, intraoperative and 10mins after operation
  heart rate, respiration rate
vital signs change | baseline, intraoperative and 10mins after operation
  respiration rate
vital signs change | baseline, intraoperative and 10mins after operation
  blood oxygen saturation of artery blood of finger(SpO2)
vital signs change | baseline, intraoperative and 10mins after operation
  mean blood pressure
vital signs change | baseline, intraoperative and 10mins after operation
  Critical-Care Observation Tool(CPOT)
vital signs change | baseline, intraoperative and 10mins after operation
  Richmond Agitation-Sedation Scale(RASS)

SECONDARY OUTCOMES:
number of adverse reaction | baseline,intraoperative,10mins after operation,30mins after operation
  respiratory depression,skeletal muscle stiffness,nausea vomting and dizziness,hypertension,allergy,bradycardia etc.

REFERENCES:
- [Result] Evane TN, Park GR. Remifentanil in the critically ill. Anaesthesia. 1997 Aug;52(8):800-1. No abstract available. PMID 9291773
- [Result] Soltesz S, Biedler A, Silomon M, Schopflin I, Molter GP. Recovery after remifentanil and sufentanil for analgesia and sedation of mechanically ventilated patients after trauma or major surgery. Br J Anaesth. 2001 Jun;86(6):763-8. doi: 10.1093/bja/86.6.763. PMID 11573581
- [Result] Wilhelm W, Dorscheid E, Schlaich N, Niederprum P, Deller D. [The use of remifentanil in critically ill patients. Clinical findings and early experience]. Anaesthesist. 1999 Sep;48(9):625-9. doi: 10.1007/s001010050762. German. PMID 10525595
- [Result] Wilhelm W, Kreuer S. The place for short-acting opioids: special emphasis on remifentanil. Crit Care. 2008;12 Suppl 3(Suppl 3):S5. doi: 10.1186/cc6152. Epub 2008 May 14. PMID 18495056
- [Result] Casey E, Lane A, Kuriakose D, McGeary S, Hayes N, Phelan D, Buggy D. Bolus remifentanil for chest drain removal in ICU: a randomized double-blind comparison of three modes of analgesia in post-cardiac surgical patients. Intensive Care Med. 2010 Aug;36(8):1380-5. doi: 10.1007/s00134-010-1836-2. Epub 2010 Mar 18. PMID 20237760
- [Result] Chalumeau-Lemoine L, Stoclin A, Billard V, Laplanche A, Raynard B, Blot F. Flexible fiberoptic bronchoscopy and remifentanil target-controlled infusion in ICU: a preliminary study. Intensive Care Med. 2013 Jan;39(1):53-8. doi: 10.1007/s00134-012-2697-7. Epub 2012 Sep 28. PMID 23052952
- [Result] Al MJ, Hakkaart L, Tan SS, Bakker J. Cost-consequence analysis of remifentanil-based analgo-sedation vs. conventional analgesia and sedation for patients on mechanical ventilation in the Netherlands. Crit Care. 2010;14(6):R195. doi: 10.1186/cc9313. Epub 2010 Nov 1. PMID 21040558
- [Result] Futier E, Chanques G, Cayot Constantin S, Vernis L, Barres A, Guerin R, Chartier C, Perbet S, Petit A, Jabaudon M, Bazin JE, Constantin JM. Influence of opioid choice on mechanical ventilation duration and ICU length of stay. Minerva Anestesiol. 2012 Jan;78(1):46-53. Epub 2011 Nov 5. PMID 21971434
- [Result] Battershill AJ, Keating GM. Remifentanil : a review of its analgesic and sedative use in the intensive care unit. Drugs. 2006;66(3):365-85. doi: 10.2165/00003495-200666030-00013. PMID 16526829
- [Result] Karabinis A, Mandragos K, Stergiopoulos S, Komnos A, Soukup J, Speelberg B, Kirkham AJ. Safety and efficacy of analgesia-based sedation with remifentanil versus standard hypnotic-based regimens in intensive care unit patients with brain injuries: a randomised, controlled trial [ISRCTN50308308]. Crit Care. 2004 Aug;8(4):R268-80. doi: 10.1186/cc2896. Epub 2004 Jun 28. PMID 15312228